CLINICAL TRIAL: NCT00407784
Title: Aldosterone-Renin Ratio to Diagnose Primary Aldosteronism in a Population of Patients With Therapy-Resistant Hypertension: Test Characteristics, Diagnostic Value and Predictive Value for Antihypertensive Treatment. The Dutch ARRAT Study.
Brief Title: Diagnostic Properties of Aldosterone-Renin Ratio in Primary Aldosteronism Among Hypertensives.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other); Pfizer (Industry)
Other Study IDs: MEC-2006-103; C05.2151; EudraCT nr: 2006-006618-13
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Hyperaldosteronism; Hypertension
Keywords: primary aldosteronism; hypertension; aldosteron-renin ratio; eplerenone; aldosteron-receptor antagonist; screening
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — Eplerenone

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: eplerenone

SUMMARY:
This study aims to evaluate the diagnostic value of the Aldosterone-Renin Ratio (ARR)as a screening test for primary aldosteronism among hypertensives. The test characteristics will be studied. Furthermore, the effect of eplerenone, a selective aldosterone-receptor antagonist will be studied.

DETAILED DESCRIPTION:
Although primary aldosteronism (PA) was formerly seen as a rare cause of hypertension, this condition is now thought to be the commonest cause of secondary hypertension, with the prevalence ranging up to 10-15 % of all hypertensives. Identification of patients with PA allows for specific treatment, for instance unilateral adrenalectomy in case of an aldosterone-producing adenoma or the administration of an aldosterone-receptor antagonist in case of bilateral adrenal hyperplasia.

Since the introduction of the aldosterone-renin ratio (ARR) as a screening tool for PA in 1981, there has been considerable debate about the diagnostic value. The values for aldosterone and renin are highly dependent on many factors, including posture, time of day and medication. Also, the cut-off values for the identification of PA remain controversial.

This study aims to evaluate the test characteristics of the ARR in a population of patients with therapy-resistant hypertension, the dependence of the ARR on medication type and the predictive value on the response on eplerenone, a selective aldosterone-receptor antagonist.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* blood pressure above 140 mmHg systolic and above 90 mmHg diastolic
* use of at least 2 antihypertensive drugs

Exclusion Criteria:

* known cause of hypertension, including white-coat hypertension
* severe renal failure (kreat > 200 umol/l)
* BMI above 32 kg/m2
* poorly regulated diabetes mellitus (HbA1C > 8.0 %)
* heart failure
* stroke or myocardial infarction within 6 months before inclusion
* angina pectoris
* pregnancy
* neoplastic disease, within 5 years before inclusion
* alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2007-01; Study Completion 2009-11

CONTACTS AND LOCATIONS:
Overall Officials: A.H. van den Meiracker, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (13):
- Netherlands (13):
  - Academical Medical Center, Amsterdam
  - VU medical Center, Amsterdam
  - IJsselland Hospital, Capelle aan den IJssel
  - Beatrix Hospital, Gorinchem
  - University Medical Center St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Ikazia Hospital, Rotterdam
  - MCRZ, lokation Zuider/Clara, Rotterdam
  - Oogziekenhuis, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - Vlietland Hospital, Schiedam
  - Ruwaard van Putten Hospital, Spijkenisse
  - Twee Steden Ziekenhuis, Waalwijk

REFERENCES:
- [Background] Hiramatsu K, Yamada T, Yukimura Y, Komiya I, Ichikawa K, Ishihara M, Nagata H, Izumiyama T. A screening test to identify aldosterone-producing adenoma by measuring plasma renin activity. Results in hypertensive patients. Arch Intern Med. 1981 Nov;141(12):1589-93. PMID 7030245
- [Background] Gordon RD, Klemm SA, Stowasser M, Tunny TJ, Storie WJ, Rutherford JC. How common is primary aldosteronism? Is it the most frequent cause of curable hypertension? J Hypertens Suppl. 1993 Dec;11(5):S310-1. No abstract available. PMID 8158400
- [Background] Strauch B, Zelinka T, Hampf M, Bernhardt R, Widimsky J Jr. Prevalence of primary hyperaldosteronism in moderate to severe hypertension in the Central Europe region. J Hum Hypertens. 2003 May;17(5):349-52. doi: 10.1038/sj.jhh.1001554. PMID 12756408
- [Background] Stowasser M, Gordon RD, Gunasekera TG, Cowley DC, Ward G, Archibald C, Smithers BM. High rate of detection of primary aldosteronism, including surgically treatable forms, after 'non-selective' screening of hypertensive patients. J Hypertens. 2003 Nov;21(11):2149-57. doi: 10.1097/00004872-200311000-00025. PMID 14597859
- [Background] Schwartz GL, Turner ST. Screening for primary aldosteronism in essential hypertension: diagnostic accuracy of the ratio of plasma aldosterone concentration to plasma renin activity. Clin Chem. 2005 Feb;51(2):386-94. doi: 10.1373/clinchem.2004.041780. PMID 15681560
- [Background] Giacchetti G, Ronconi V, Lucarelli G, Boscaro M, Mantero F. Analysis of screening and confirmatory tests in the diagnosis of primary aldosteronism: need for a standardized protocol. J Hypertens. 2006 Apr;24(4):737-45. doi: 10.1097/01.hjh.0000217857.20241.0f. PMID 16531803
- [Background] Kaplan NM. The current epidemic of primary aldosteronism: causes and consequences. J Hypertens. 2004 May;22(5):863-9. doi: 10.1097/00004872-200405000-00001. PMID 15097219